CLINICAL TRIAL: NCT05596123
Title: Therapeutic Chinese Foot Massage for Peripheral Neuropathy Symptoms Among People With Human Immunodeficiency Virus: A a Randomized Controlled Trial
Brief Title: Tui na for Peripheral Neuropathy Among People With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston Downtown (Other)
Responsible Party: Principal Investigator, Song Ge, Assistant Professor, University of Houston Downtown
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UHDowntown
Record Dates: First submitted 2022-10-17; First posted 2022-10-27 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a prospective, two-arm, double-blinded, randomized controlled trial. A one-to-one ratio will be used to randomly assign participants to the TCFM group or the placebo massage group. Six weekly 25-minute TCFM sessions will be delivered to participants in the TCFM group. Six weekly 25-minute sessions of placebo massage will be delivered to participants in the placebo massage group.
Who Masked: Participant, Investigator
Masking Description: Participants, the outcome assessors, and the statistician will be unaware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- therapeutic Chinese foot massage (TCFM) (Experimental): A one-to-one ratio will be used to randomly assign participants to the TCFM group or the placebo massage group.
  Interventions: Behavioral: Therapeutic Chinese foot massage
- The Placebo Massage Group (Placebo Comparator): Six weekly 25-minute TCFM sessions will be delivered to participants in the TCFM group.
  Interventions: Behavioral: Placebo massage

INTERVENTIONS:
Behavioral: Therapeutic Chinese foot massage — Participants in the TCFM group will receive six weekly 25-minute TCFM sessions by a therapist. Each session will start with an assessment of the legs and toes of the affected extremity for broken skin and lesions, which the therapist will try to avoid. The participant will be positioned with support to their foot and legs, with the sole directed downward and the therapist directly in alignment with the soles of the foot. The therapist will sequentially perform the following four steps for each TCFM session.
  Arms: therapeutic Chinese foot massage (TCFM)
Behavioral: Placebo massage — The same therapist will give six weekly 25-minute placebo massage sessions to participants in the placebo massage group. These sessions will include assessing the affected extremity's legs and toes for lesions and broken skin in order to avoid them during the massage, as well as gentle foot and toe rubbing without any point stimulation or other TCFM techniques.
  Arms: The Placebo Massage Group

SUMMARY:
Peripheral neuropathy (PN) is a common neurological complication in people with human immunodeficiency virus (PHIV) with no Food and Drug Administration-approved treatment. Medications commonly used to treat HIV-related PN are not effective and have many side effects. HIV-related PN symptoms may be alleviated or treated with therapeutic Chinese foot massage (TCFM), a non-invasive, relatively safe, non-pharmacological intervention.

DETAILED DESCRIPTION:
This is a prospective, two-arm, double-blinded, randomized controlled trial. Aim: This trial aims to assess the effectiveness of TCFM on HIV-related PN in people with HIV (PHIV).

ELIGIBILITY:
Inclusion Criteria:

1. have confirmed HIV diagnosis
2. self-report PN-related symptoms in their lower extremity, such as sharp, jabbing, throbbing, or burning pain, numbness, decreased sensation to pinprick, prickling or tingling feeling, lack of coordination and falling muscle weakness, and extreme sensitivity to touch
3. are not taking any medications, including pain medicine, to alleviate PN
4. age 18 years and older
5. can communicate with researchers in English or Mandarin Chinese
6. are not pregnant or lactating
7. are not concurrently enrolled in other clinical trials.

Exclusion Criteria:

1) People who have received any non-pharmacological interventions, including massage to treat their PN symptoms in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Lower extremity pain | at 6 months
  The numeric pain scale has a score range between 0 and 10. A higher score indicates more pain.
Lower extremity functioning | at 6 months
  The lower extremity functioning scale has a score range between 0 and 80. A higher score indicates better functioning.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Ge S, Dune L, Yang C, Tian C, Wang Y. Tui Na for painful peripheral neuropathy in people with human immunodeficiency virus: A randomized, double-blind, placebo-controlled trial protocol. Front Neurol. 2023 Feb 23;14:1113834. doi: 10.3389/fneur.2023.1113834. eCollection 2023. PMID 36908633